CLINICAL TRIAL: NCT01108367
Title: Predictor of Transient Urinary Incontinence Following Holmium Laser Enucleation of the Prostate
Brief Title: Transient Urinary Incontinence After Holmium Laser Enucleation of the Prostate (HoLEP)
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Seung Paick/M.D.,Ph.D., Seoul National University Hospital
Other Study IDs: HoLEPUI
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Prostatic Hyperplasia; Incontinence
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
In men, urinary incontinence (UI) is relatively uncommon, and usually associated with some forms of prostate surgery. Thus, one of the risks of surgery for benign prostate hyperplasia (BPH) is postoperative UI. The guidelines of the American Urological Association for BPH treatment indicate that UI (2~5%) is relevant complications after transurethral prostatectomy (TURP). Rassweiler et al., based on a review of publications stated that early UI may occur in up to 30-40% of patients after TURP. Rigatti et al. reported that early postoperative urgency UI occurred in 38.6% (TURP) and 44% (holmium laser enucleation of the prostate; HoLEP) of surgically treated patients at 1-month after the surgery. Recently, the follow-up data for patients treated with HoLEP showed that transient stress UI developed in up to 44% after HoLEP. Although this alternative surgical treatment such as HoLEP can be performed safely with minimal complications, patients often face debilitating UI during the postoperative period before any improvement in micturition parameters occurs. Although this symptom ameliorates within a relatively short time, it usually cause significant stress and anxiety to the patient as far as their durations is concerned. In addition to its economic cost, UI is a distressing condition that has major impacts on a patient's quality of life. Social withdrawal, isolation, and depression occur in some patients.

Because this problem is usually temporary, there has been little attempt at addressing the issue. Therefore, there has been no research devoted specifically to transient de novo UI associated with HoLEP.

1. The aim of the present study was following:

1. to investigate the incidence of transient de novo UI after HoLEP for BPH
2. determine the predictors of early postoperative transient de novo UI.

ELIGIBILITY:
Inclusion Criteria:

* age older than 50 years
* presence of moderate or severe LUTS (International Prostate Symptom Score [IPSS] greater than 8)or maximum flow rate of less than 10 mL/s

Exclusion Criteria:

* previous prostate surgery
* urethral stricture
* prostate carcinoma
* neurogenic bladder disease

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men who underwent HoLEP for lower urinary tract symptoms (LUTS) with BPH refractory to alpha blocker medication
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Cho, M.D., Principal Investigator — Seoul National University Hospital; Jae-Seung Paick, M.D.,Ph.D., Study Chair — Seoul National University Hospital

REFERENCES:
- [Result] Cho MC, Park JH, Jeong MS, Yi JS, Ku JH, Oh SJ, Kim SW, Paick JS. Predictor of de novo urinary incontinence following holmium laser enucleation of the prostate. Neurourol Urodyn. 2011 Sep;30(7):1343-9. doi: 10.1002/nau.21050. Epub 2011 Apr 28. PMID 21538499